CLINICAL TRIAL: NCT01172015
Title: NK-ITP STUDY : NATURAL KILLER CELLS IN IMMUNOLOGIC THROMBOCYTOPENIC PURPURA OF ADULTS.
Brief Title: NATURAL KILLER CELLS IN IMMUNOLOGIC THROMBOCYTOPENIC PURpura of Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010-A00396-33; 2010 03 (Other: ap hm)
Record Dates: First submitted 2010-07-26; First posted 2010-07-29 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Immunologic Thrombcytopenic Purpura (ITP) Adults
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTI patients (Experimental): Study NK cells functions, phenotypic changes and transcripts from ITP patients
  Interventions: Other: blood samples
- healthy volunteers (Other): Study NK cells functions, phenotypic changes and transcripts from healthy volunteers
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples

SUMMARY:
Immunologic thrombcytopenic purpura (ITP) affects both children and adults. The incidence is estimated in adults about 1,6/100 000/per year. Chronic and relapsing forms of the disease that represent 70% of adult cases are associated with impairment of quality of life related to treatments side effects and bleeding. ITP is secondary to the destruction of circulating platelets through an auto-immune process and to a decrease of platelet production in bone marrow. Auto antibodies are usually directed against epitopes of the GPIIb/IIIa, expressed by platelets. The destruction of the platelets seems to occur mainly in the spleen through antibody dependent cytotoxicity. Both macrophages and cytotoxic T lymphocytes subsets participate to the platelet destruction through the CD16, the low affinity receptor for the Fc of IgG. Thus the CD16 "pathway" is a target for treatments in ITP as for example intravenous immunoglobulins and more recently inhibitors of the syk kinase.

DETAILED DESCRIPTION:
Natural Killer cells (NK) cells, who are now implicated in the pathophysiology of several autoimmune diseases, express CD16 and display antibody dependent cytotoxicty. Moreover NK cells are present in human spleen. However their role in ITP has not been studied so far. NK could represent a new target for treatments in ITP. We propose thus to conduct a study to characterizes NK cells changes in patients with ITP.

ELIGIBILITY:
Inclusion Criteria:

* ITP patients,platelets less than 50000 G/L

Exclusion Criteria:

* Secondary ITP (VIH, VHC...)
* treatment with Immunosuppressive agents except corticoids (10 mg/day)
* treatment with Ig IV less than 3 weeks
* treatment with Rifuximab less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Compare NK cells functions, phenotypic changes and transcripts from ITP patients and controls in a case control, multicentric study | 24 months
  Flow cytometry,transcripts.

SECONDARY OUTCOMES:
Influence of the Ig (IV) treatment on ITP patients' NK cells | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Schleinitz Nicolas, Principal Investigator — APHM
Locations (1):
- APHM, Marseille, France